CLINICAL TRIAL: NCT07216534
Title: Piloting a Virtual Reality-Based, Randomized Controlled Trial of Psychosocial Responses to Neighborhood Physical Disorder
Brief Title: Virtual Reality Viewing of Unaltered Streetscape Versus Digitally Manipulated Opposite Streetscape to Assess Psychosocial Response in Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jesse Plascak, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-25170; NCI-2025-07331 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm; Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (twin followed by opposite streetscape) (Experimental): Participants have their streetscape photographed. Participants view a standard residential streetscape using VR for up to 5 minutes. Patients then view a digital twin of their streetscape with identical physical disorder using VR for up to 5 minutes followed by viewing their streetscape with the opposite physical disorder using VR for up to 5 minutes.
  Interventions: Other: Survey Administration; Other: Virtual Technology Intervention
- Arm II (opposite followed by twin streetscape) (Experimental): Participants have their streetscape photographed. Participants view a standard residential streetscape using VR for up to 5 minutes. Patients then view their streetscape with the opposite physical disorder using VR for up to 5 minutes followed by viewing a digital twin of their streetscape with identical physical disorder using VR for up to 5 minutes.
  Interventions: Other: Survey Administration; Other: Virtual Technology Intervention

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Other: Virtual Technology Intervention — View standard streetscape
  Other Names: Virtual Reality Intervention; Virtual Technology
Other: Virtual Technology Intervention — View digital twin of streetscape
  Other Names: Virtual Reality Intervention; Virtual Technology
Other: Virtual Technology Intervention — View opposite digital streetscape
  Other Names: Virtual Reality Intervention; Virtual Technology

SUMMARY:
This clinical trial compares virtual reality viewing of an unaltered streetscape versus a digitally manipulated opposite streetscape to assess the psychosocial response in participants. Visible measures of neighborhood factors might be associated with health outcomes and risk factors of those outcomes. Short-term exposure to virtual reality environments representing very high or very low levels of neighborhood physical disorder - presence or absence of garbage/litter, presence or absence of graffiti, presence or absence of an abandoned building, presence or absence of large dumpsters, poor or very well-kept building conditions, poor or very well-kept yard conditions, poor or very well-kept road verge conditions may be a safe and effective way to assess psychosocial response in participants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare sympathetic autonomic measures (heart rate variability and skin conductance) between participants viewing, in virtual reality, their streetscape as a digitally manipulated opposite version with respect to physical disorder indicators versus participants viewing their streetscape as a digital twin with respect to physical disorder indicators.

II. Compare self-report measures (Self-Assessment Manikin and state anxiety ratings) between participants viewing, in virtual reality, their streetscape as a digitally manipulated opposite version with respect to physical disorder indicators versus participants viewing their streetscape as a digital twin with respect to physical disorder indicators.

III. Record side effects of interacting within a virtual reality environment over short periods of time (3-5 min):

IIIa. Quantify frequency of side effects; IIIb. Explore whether side effects increase across subsequent VR sessions of the cross-over study; IIIc. Explore whether side effects vary by VR intervention arm (digital twin of own streetscape or digitally manipulated opposite indicators of physical disorder of own streetscape).

IV. Analyze impact of covariates on study outcomes.

EXPLORATORY OBJECTIVES:

I. Compare eye gaze density between participants viewing, in virtual reality, their streetscape as a digitally manipulated opposite version with respect to physical disorder indicators versus participants viewing their streetscape as a digital twin with respect to physical disorder indicators.

II. Compare self-report measures (neighborhood social cohesion and neighborhood disorder) between participants viewing, in virtual reality, their streetscape as a digitally manipulated opposite version with respect to physical disorder indicators versus participants viewing their streetscape as a digital twin with respect to physical disorder indicators.

OUTLINE: Participants are randomized within their residing neighborhood to 1 of 2 arms.

ARM I: Participants have their streetscape photographed. Participants view a standard residential streetscape using virtual reality (VR) for up to 5 minutes. Patients then view a digital twin of their streetscape with identical physical disorder using VR for up to 5 minutes followed by viewing their streetscape with the opposite physical disorder using VR for up to 5 minutes.

ARM II: Participants have their streetscape photographed. Participants view a standard residential streetscape using VR for up to 5 minutes. Patients then view their streetscape with the opposite physical disorder using VR for up to 5 minutes followed by viewing a digital twin of their streetscape with identical physical disorder using VR for up to 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+
* Must currently live (4+ night/week) at the residence being studied. Only one resident per household will be selected
* Must understand and be able to read English
* Must agree to have residence photographed
* Must be able to wear a VR head mounted display
* Must live in neighborhood that has been selected for study
* Must be willing and able to attend an approximately 2 hour in-person visit on Ohio State University (OSU) campus

Exclusion Criteria:

* Pregnant women
* Visual or mobility impairment
* Cannot have epilepsy or other condition that would inhibit them from being able to use a VR headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability | From baseline to completion of virtual reality (VR) viewings, up to 1 day
  Mean heart rate variability over the entire session of each VR condition will be calculated from electrocardiograph data. Will compare the difference between two VR conditions (viewing opposite neighborhood image versus viewing twin neighborhood image) using a crossover design. Analyses of outcomes will be conducted using generalized linear mixed model approaches.
Change in skin conductance | From baseline to completion of VR viewings, up to 1 day
  Skin conductance, measured as microsiemens, will be calculated as the mean value over each VR condition. Will compare the difference between two VR conditions (viewing opposite neighborhood image versus viewing twin neighborhood image) using a crossover design. Analyses of outcomes will be conducted using generalized linear mixed model approaches.
Affective reaction | After completion of VR viewings, up to 1 day
  Assessed via Self-assessment Manikin. Will compare the difference between two VR conditions (viewing opposite neighborhood image versus viewing twin neighborhood image) using a crossover design. Analyses of outcomes will be conducted using generalized linear mixed model approaches.
Anxiety | After completion of VR viewings, up to 1 day
  Assessed via Spielberger State-Trait Anxiety Inventory short form. Will compare the difference between two VR conditions (viewing opposite neighborhood image versus viewing twin neighborhood image) using a crossover design. Analyses of outcomes will be conducted using generalized linear mixed model approaches.
Participant reported discomfort | After completion of VR viewings, up to 1 day
  This is an open-ended outcome measure. Discomfort reported by participants will be recorded by study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Plascak, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu